CLINICAL TRIAL: NCT03357237
Title: RANDOMIZED, DOUBLE-BLIND CLINICAL TRIAL TO EVALUATE EFFICACY AND SAFETY OF XILOGLUCAN IN ACUTE GASTROENTERITIS IN CHILDREN
Brief Title: EFFICACY AND SAFETY OF XILOGLUCAN IN ACUTE GASTROENTERITIS IN CHILDREN
Acronym: PEDXIL01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Enriqueta Roamn (Other)
Responsible Party: Sponsor-Investigator, Enriqueta Roamn, MD, Puerta de Hierro University Hospital
Organization: Puerta de Hierro University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEDXIL 01
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: * Intervention or experimental group: treatment regimen with oral rehydration solution and xyloglucan
  * Control or reference group: treatment regimen with oral rehydration solution and placebo.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XYLOGLUCAN (Experimental): treatment regimen with oral rehydration solution and xyloglucan
  Interventions: Other: medical device
- PLACEBO (Placebo Comparator): rehydration solution and placebo.
  Interventions: Other: medical device

INTERVENTIONS:
Other: medical device — patients will be assigned, following an external randomization, to two groups:
  * Intervention or experimental group: treatment regimen with oral rehydration solution and xyloglucan
  * Control or reference group: treatment regimen with oral rehydration solution and placebo

SUMMARY:
Acute gastroenteritis (GEA) is an inflammation of the intestinal mucosa that clinically translates into an acute episode of diarrhea and vomiting and is generally associated with an intestinal infectious disease. It is one of the most common diseases in children and an important cause of morbidity and mortality worldwide. The important loss of liquids can lead to dehydration, acidosis and hydroelectrolitic alteration. Infants are more vulnerable to gastrointestinal infection and its consequences, dehydration and malnutrition.

There is no specific treatment, so it is exclusively symptomatic

A new type of products considered as mucoprotectors has been developed, such as gelatin tannate or xyloglucan, still with little data to establish recommendations on its use in the GEA. They would be able to reproduce in the intestine a muco-adhesive film or sheet protective It must be considered in this sense that mucus is the first barrier that protects the gastrointestinal tract against microorganisms or antigens and that bacterial invasion is related to the opening of narrow junctions.

Xyloglucan was approved in Europe as a medical device IIa to restore the physiological functions of the intestinal wall in the form of capsules for adults and envelopes for children.

DETAILED DESCRIPTION:
A randomized, blinded study with a control group is proposed in this project to establish solidly the efficacy of xyloglucan in the treatment of acute gastroenteritis in children.

The main variable of evaluation will be the duration of diarrhea, defined as the time it takes to normalize the consistency of stools (according to the Bristol or Amsterdam scale) or their number.

Clinical trial in phase IV with medical product type IIa and CE marking, used in the same conditions in which it is marketed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical of acute gastroenteritis: change in the consistency of stools to "loose" or liquid according to Bristol scale (6 or 7) or Amsterdam (infants) (A) and / or increase in the number of stools (greater or equal to 3 / day) with a duration of less than 72 h
* Age over 3 months and under 5 years
* Written informed consent according to ICH / GCP and local legislation, obtained before any study procedure of parents or guardians

Exclusion Criteria:

* Treatment with antibiotics, xyloglucan, gelatin tannate, racecadotril, smectite, probiotics or zinc (including oral rehydration solution containing zinc and / or probiotics) in the previous week
* Exclusive breastfeeding
* Chronic gastrointestinal disease (celiac disease, cystic fibrosis, inflammatory bowel disease, food allergy)
* Immunodeficiencies
* Malnutrition (weight / height / length less than P3 according to WHO standards)
* Severe dehydration
* Impossibility of follow-up
* Known hypersensitivity to gelatin or xyloglucan
* Absence of informed consent
* Caregivers / parents who can not understand or comply with all the instructions and requirements of the study.
* If in the opinion of the researcher there are findings in the physical examination, abnormalities in the results of the clinical analyzes or other medical, social or psychosocial factors that could negatively influence

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
time of resolution of diarrhea | 14 days
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Enriqueta Roman, PHD, Study Director — Hospital Universitario Puerta de Hierro Majadahonda
Locations (1):
- Hospital Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided